CLINICAL TRIAL: NCT06814158
Title: A Phase II Study of Neoadjuvant Ivonescimab Combined with Chemotherapy in Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant Ivonescimab and Chemotherapy in Resectable Esophageal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Hongjing Jiang, Director of Department Esophageal Surgery, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E20241631A; E20241631A (Other: Tianjin Medical University Cancer Institute and Hospital)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Esophageal Squamour Cell Cancer
Keywords: Esophageal cancer; Squamous cell carcinoma; Neoadjuvant therpay; VEGF-A; PD-1; Immunotherapy; Ivonescimab
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Squamous Cell | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Ivonescimab Combined with Chemotherapy (Experimental): Ivonescimab 20mg/kg + chemotherapy (Cisplatin + Paclitaxel) Q3W, 3 cycles
  Interventions: Drug: Ivonescimab Combined With Chemotherapy

INTERVENTIONS:
Drug: Ivonescimab Combined With Chemotherapy — Ivonescimab 20mg/kg + CT Q3W, 3cycles

SUMMARY:
Neoadjuvant ChemoRadioTherapy (NCRT) combined with surgical resection is the standard treatment for locally advanced esophageal squamous cell carcinoma (ESCC) based on CROSS and 5010 study. However, the recurrence and metastasis rate after neoadjuvant therapy is still very high, reaching about 40%, which seriously affects the long-term survival of patients after surgery. Therefore, how to improve the neoadjuvant therapy regimen, thereby increasing the pCR rate of ESCC patients, eliminating micro metastases and prolonging survival, has always been an urgent problem to be solved in clinical practice. The combination of neoadjuvant chemotherapy and immunotherapy significantly improved the perioperative outcomes of ESCC patients, and the safety and efficacy of the chemoimmunotherapy were validated in the population of locally advanced ESCC patients (Keystone 001 and ESCORT-NEO study). The Ivonescimab Injection is an IgG1 subtype humanized bispecific antibody that targets human vascular endothelial growth factor-A (VEGF-A) and programmed death protein-1 (PD-1). It can simultaneously bind to VEGF-A and PD-1, competitively block the interaction between VEGF-A, PD-1 and their ligands, and exert immune and anti angiogenic effects. This innovative antibody structure design effectively reduces the side effects and enhances the safety of the drug therapy. A few clinical trials (HARMONi-A and HARMONi-2study) suggest that the combination therapy of Ivonescimab and chemotherapy for locally advanced ESCC may be safe and effective, and is expected to achieve better therapeutic effects than neoadjuvant chemoimmotherapy. This study aims to explore the safety and efficacy of Ivonescimab combination with chemotherapy in the treatment of locally advanced resectable ESCC (cII-III stage), and analyze the feasibility of this treatment regimen. At the same time, a comprehensive analysis and detection of the tumor immune microenvironment, circulating immune cells, and circulating tumor DNA (ctDNA) in ESCC were conducted to elucidate the role of immune status and dynamic changes in ctDNA for predicting therapeutic efficacy and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* 1) Histologically confirmed primary esophageal squamous cell carcinoma, locally advanced, staging cT1N2M0, cT2-3N0-2M0 (stage II/III), AJCC 8th edition clinical staging of esophageal squamous cell carcinoma; 2) Surgical treatment is possible; 3) ECOG score: 0 to 1; 4) The function of important organs meets the following requirements (excluding the use of any blood components and cell growth factors within 14 days): the subject has no dysfunction of major organs, and the blood routine, lung, liver, kidney function, and heart function are basically normal. Laboratory laboratory test indicators must meet the following requirements: blood: white blood cells>4.0 × 109/L, absolute count of neutrophils (ANC) ≥ 2.0 × 109/L, platelet count>100 × 109/L, hemoglobin>90g/L; Pulmonary function: FEV1 ≥ 1.2L, FEV1% ≥ 50%, and DLCO ≥ 50%; Liver function: serum bilirubin is below 1.5 times the maximum normal value; ALT and AST are 1.5 times lower than the maximum normal values. Renal function: Blood creatinine (SCr) ≤ 120 µ mol/L, creatinine clearance rate (CCr) ≥ 60 ml/min; 5) Before treatment, gastroscopy tissue and blood samples need to be collected from our center; 6) The subjects voluntarily joined this study, showed good compliance, and cooperated with safety and survival follow-up.

Exclusion Criteria:

* 1) Previously received radiation therapy, chemotherapy, hormone therapy, surgery, or molecular targeted therapy; 2) Suspected cervical lymph node metastasis on imaging; The subject has a history or concurrent history of other malignant tumors (Excluding cured basal cell carcinoma of the skin and cervical carcinoma in situ; 3) Previous PD-1/PD-L1 treatment history; 4) History of allergies to macromolecular protein preparations or any PD-1 components; 5) Subjects with any active autoimmune disease or history of autoimmune disease (such as but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or complete remission of childhood asthma without any intervention in adulthood; subjects with asthma requiring medical intervention with bronchodilators cannot be included); 6) The subject is currently using immunosuppressive agents, systemic or absorbable local hormone therapy to achieve immunosuppressive effects (dose>10mg/day prednisone or other therapeutic hormones), and has continued to use them within 2 weeks prior to enrollment; 7) Ascites or pleural effusion with clinical symptoms require therapeutic puncture or drainage; 8) Patients with uncontrolled cardiac clinical symptoms or diseases, such as: (1) NYHA grade 2 or above heart failure, (2) unstable angina, (3) myocardial infarction within 1 year, and (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; 9) Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg>2g/L), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy; 10) The patient currently (within 3 months) has digestive tract diseases such as esophageal varices, active ulcers in the stomach and duodenum, ulcerative colitis, portal hypertension, or active bleeding from unresected tumors, or other conditions determined by the researchers that may cause gastrointestinal bleeding or perforation; 11) Previous or current severe bleeding (bleeding>30 ml within 3 months), hemoptysis (fresh blood >5ml within 4 weeks) or thromboembolic events (including stroke events and/or transient ischemic attacks) occurring within 12 months; 12) The subject has an active infection or an unexplained fever >38.5℃ during the screening period or before the first administration (according to the researcher's judgment, subjects with fever caused by tumors can be included in the group); 13) Having experienced abdominal fistula, gastrointestinal perforation, or abdominal abscess less than 4 weeks prior to medication; 14) Patients with objective evidence of past and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe impairment of lung function, etc; 15) Subjects with congenital or acquired immune function defects, such as HIV infection, or active hepatitis (transaminase does not meet the inclusion criteria, hepatitis B reference: HBV DNA ≥10^4/ml ； Hepatitis C reference: HCVRNA≥10^3/ml）； Chronic hepatitis B virus carriers with HBV DNA<2000 IU/ml (<10^4 copies/ml) must receive antiviral treatment during the trial period in order to be enrolled; 16) The subjects are currently participating in other clinical studies or have been less than one month since the end of the previous clinical study; Participants may receive other systemic anti-tumor treatments during the study period; 17) Medication less than 4 weeks before the study or may receive live vaccine during the study period; 18) The subject is known to have a history of substance abuse, alcoholism, or drug use; 19) The subject is unable or unwilling to bear the self funded portion of the examination and treatment costs; 20) The researchers believe that the subjects should be excluded from this study, for example, if the researchers determine that there are other factors that may cause the study to be terminated midway, such as other serious illnesses (including mental illnesses) that require concomitant treatment, serious laboratory abnormalities, accompanied by family or social factors, which may affect the safety of the subjects, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response, pCR | From enrollment to the postoperative pathology report at 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Hospital, Hexi District, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
IPD will be shared based on the request from other researchers.